CLINICAL TRIAL: NCT04982692
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase Ⅲ, Efficacy and Safety Study of INTRAROSA® (Prasterone) Vaginal Inserts on Postmenopausal Vulvovaginal Atrophy (VVA)
Brief Title: A Clinical Study of INTRAROSA® (Prasterone) Vaginal Inserts in Postmenopausal Vulvovaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INT-ZK-2021
Record Dates: First submitted 2021-06-23; First posted 2021-07-29 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Postmenopausal Vulvovaginal Atrophy
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravaginal prasterone (Experimental): 6.5 mg of Intravaginal prasterone once daily at bedtime with a finger to insert the vaginal suppository into the vagina for a treatment cycle of 12 weeks.
  Interventions: Drug: intravaginal prasterone
- Placebo ovules (Placebo Comparator): Placebo ovules once daily at bedtime with a finger to insert the vaginal suppository into the vagina for a treatment cycle of 12 weeks.
  Interventions: Drug: Placebo ovules

INTERVENTIONS:
Drug: intravaginal prasterone — 6.5 mg of Intravaginal prasterone once daily at bedtime with a finger to insert the vaginal suppository into the vagina for a treatment cycle of 12 weeks.
  Other Names: Intrarosa
  Arms: Intravaginal prasterone
Drug: Placebo ovules — Placebo ovules once daily at bedtime with a finger to insert the vaginal suppository into the vagina for a treatment cycle of 12 weeks.
  Arms: Placebo ovules

SUMMARY:
This study is a phase III which includes two treatment phases. The phase 1 study is a multi-center, randomized, double-blind, placebo- controlled, parallel group that provide primary efficacy and safety data.

The Phase 2 study is a single-arm, open-label conducted in a subset of subjects who completed the phase 1 study to provid additional long-term safety and efficacy.

DETAILED DESCRIPTION:
The phase 1 study which includes the screening phase (up to 3 weeks) and treatment phase (12 weeks). After signing the informed consent, the inclusion and exclusion criteria will be confirmed preliminarily at screening visit and reconfirmed at Day 1 (baseline). At least 418 eligible subjects will be randomized in a 1:1 ratio to receive 6.5mg of intravaginal prasterone or placebo once-daily for 12 weeks.

The phase 2 study which includes the treatment phase (26 weeks). A total of 100 subjects who have completed Phase 1, not occur adverse event（AE） grade ≥3 or serious adverse event (SAE), or recover all AE grades ≤1, and voluntary to participate in Phase 2 study. After signing the ICF, the subject will receive 6.5mg of intravaginal for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 40 and 80 years of age inclusive;
2. Menopausal women (with or without hysterectomy) must also meet 1 of the following 3 conditions:

   A Non-hysterectomy, menopause ≥ 12 months; B. Menopause > 6 months and < 12 months or premenopausal hysterectomy, follicle stimulating hormone (FSH) > 40 IU/L; C ≥ 6 months since baseline assessment (Day 1) with or without hysterectomy.
3. At screening and baseline (Day 1), the subject presented with moderate-severe dyspareunia (dyspareunia) as measured by the Vaginal Atrophy Symptom Questionnaire (VASQ) and self-rated as the most bothersome symptom.
4. ≤ 5% superficial cells by vaginal smear at screening and baseline (Day 1).
5. Vaginal pH > 5 at Screening and Baseline (Day 1).
6. Women (with or without a partner) who currently have sex or other sexual activity (masturbation, etc.) at least once a month, or who have sex or other sexual activity at least once a month in the past, with reduced sexual activity due to excessive pain or vaginal dryness.
7. Normal physical examination of the breast and normal mammographic findings (BI-RADS grade 1 or 2) within 9 months prior to the baseline visit (Day 1).
8. Normal cervical smear results (including inflammatory changes), regardless of hysterectomy (no abnormal cervical smear in the past 2 years if ASCUS is present, and human papillomavirus (HPV) test negative can be used) within 12 months before the baseline visit (Day 1).
9. Voluntarily participate in this clinical trial and sign the informed consent form (ICF).

   -

Exclusion Criteria:

1. Patients with a history of malignant tumor.
2. Have active or history of thromboembolic disease (excluding thromboembolic events due to accidents, surgery, immobilization).
3. Clinically significant endocrine metabolic disease (e.g., diabetes mellitus) not controlled with medication.
4. Use of estrogen injections, estrogen implant sticks, progestogen injections, progestogen implants, androgens, anabolic steroids within 6 months of the screening visit.
5. Use oral estrogen, oral progesterone, prasterone (DHEA) or intrauterine progesterone treatment, intravaginal hormonal drugs (ring, cream, gel or tablet), estrogen alone or estrogen/pregnancy within 8 weeks before the screening visit, hormone transdermal drug users.
6. Confirmed depression with poor control under standard treatment or history of diagnosed psychiatric disorder.
7. Those who have participated in or plan to participate in other drug or device clinical trials during the study period within 1 month prior to the screening visit.
8. Laboratory findings suggestive of glutamic-pyruvic transaminase (ALT), glutamic oxaloacetic transaminase (AST) ≥ 2 times the upper limit of normal, or creatinine ≥ 1.5 times the upper limit of normal.
9. Grade 2 and higher uterine prolapse (cervix reaching labia minora).
10. Transvaginal ultrasound revealed a uterine fibroid ≥ 3 cm in diameter.
11. Endometrial thickness ≥ 4 mm by transvaginal ultrasound, or other comprehensive assessment by the investigator with the possibility of endometrial hyperplasia, deterioration.
12. Current endometrial polyps.
13. Previous endometrial ablation.
14. Patients with vulvar lichen sclerosus.
15. Patients with unexplained vaginal bleeding.
16. Patients who are known to be allergic to the study drug or its ingredients.
17. Patients who have participated in other relevant clinical trials of the investigational drug (prasterone vaginal suppositories).
18. History of past or present drug or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine).
19. Subjects who are unable to perform the procedures required by the protocol, or any other subjects who are not suitable for this clinical study judged by the investigator.

    -

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
The change in the dyspareunia (dyspareunia) severity score at Day 85. | week 12
  Compared with Day 1, the changes in the dyspareunia (dyspareunia) severity score (by VASQ) at Day 85 (12 weeks) in the two groups of subjects.
The change in the vaginal pH at Day 85. | week 12
  Compared with Day 1, the changes in the vaginal pH changes at Day 85 (12 weeks) in the two groups of subjects.
The change in the proportion of parabasal cells at Day 85. | week 12
  Compared with Day 1, the changes in the proportion of parabasal cells at Day 85 (12 weeks) in the two groups of subjects.
The change in the proportion of superficial cells at Day 85. | week 12
  Compared with Day 1, the changes in the proportion of superficial cells at Day 85 (12 weeks) in the two groups of subjects.

SECONDARY OUTCOMES:
Change in vaginal dryness and vaginal irritation/itching severity score at day 85 (12 weeks). | week 12
  Compared with the baseline period, at day 85 (12 weeks) in both groups: change in vaginal dryness and vaginal irritation/itching severity score by VASQ.
Change in Female Sexual Function Index at Day 85 (12 weeks). | week 12
  Compared with the baseline period, the two groups at Day 85 (12 weeks): change in Female Sexual Function Index (FSFI questionnaire).
Effects on DHEA in blood | week 12
  To test the concentrations of DHEA in blood.
Changes in the gynecological vaginal examination. | week 12
  The changes of total severity score in the vaginal discharge, vaginal epithelial integrity, vaginal epithelial surface thickness, and vaginal color by gynecological vaginal examination.
Adverse event. | week 6，week 12
  The proportion of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: long Sui, Principal Investigator — No. 419, Fangxie Road, Huangpu District, Shanghai
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No